CLINICAL TRIAL: NCT03879785
Title: TAPS-ESP: Tobacco, Alcohol, Prescription Drug, and Illicit Substance Use Electronic Spanish Platform
Acronym: TASP-ESP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 018-596
Record Dates: First submitted 2019-03-12; First posted 2019-03-19 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Tobacco, Alcohol, Prescription Drug, and Illicit Substance Use
Keywords: Tobacco; Alcohol; Prescription Drug; Illicit Substance Use; Screening; Spanish; Hispanic
MeSH Terms: interventions — Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Administration followed by Interviewer-Administered (Active Comparator)
  Interventions: Other: Screening
- Interviewer-Administered followed by Self-Administration (Active Comparator)
  Interventions: Other: Screening

INTERVENTIONS:
Other: Screening — Screening and validation of assessment tool translated into Spanish

SUMMARY:
This Phase 1 STTR project will develop a technology platform for delivering the TAPS Tool to a Spanish-speaking, health disparity population in a community health center. This will involve the adaptation of the TAPS into Spanish, its deployment on a self-administered mobile/tablet technology platform, and an empirical study of its preliminary validity, feasibility, and acceptability in a Spanish-speaking primary care sample. The investigators refer to this novel adaptation of the TAPS Tool as the TAPS-Electronic Spanish Platform, or TAPS-ESP.

DETAILED DESCRIPTION:
Linguistically Accurate Screening and Assessment is Critical for Quality Patient Care. Accurate screening, diagnosis and treatment are entirely dependent on a linguistically-accurate and culturally-relevant assessment, especially for sensitive topics such as substance use. Language accessibility is essential to quality healthcare, the lack of which is an independent predictor of poor control of chronic disease and a significant contributor to health disparities, lack of patient satisfaction with healthcare, and poor quality patient education and understanding of their disorder. Hispanics experience a disproportionate burden of disability associated with mental disorders because of these disparities.

Primary care settings often are the gateway to identifying undiagnosed or untreated behavioral health disorders through effective screening. Thus, primary care settings can play a critical role in reducing behavioral health disparities by identifying individuals at risk of substance use problems. As the first steps in ensuring access to appropriate intervention or linkage to treatment services, screening and assessment are essential ingredients in quality care. It is widely believed that substance use problems are over represented in primary care settings, but providers lack the tools to effectively screen. Most of the patients seen in primary care are unlikely to seek treatment in the specialty behavioral health service system. Moreover, failure to identify unhealthy alcohol and other drug use can produce harmful medication interactions, resulting in significant clinical complications.

The "Tobacco, Alcohol, Prescription medication, and illicit Substance use screening Tool (or TAPS Tool), is a two-stage screening and brief assessment tool that first screens the four broad substance abuse categories (tobacco, alcohol, prescription drug misuse, and illicit substance use). In the second stage, the patient is assessed for more specific risks related to an expanded array of substances (tobacco, alcohol, cannabis, cocaine, methamphetamines, prescription stimulants, heroin, prescription opioids, sedatives, and other substances). The 4-item screener triggers brief assessment on these substance categories, and each substance yields a score of 0-3 (except alcohol, which is scored on a 0-4 range), which conveys to providers whether an intervention is indicated (a score of 1 suggests sub-diagnostic problem use; a score of 2 suggests substance use disorder). The TAPS Tool was validated against established diagnostic assessments in both interviewer-administered and self-administered iPad formats in a large, multi-site study (described in Preliminary Studies, below). However, only 11.7% of the original TAPS study sample reported Hispanic ethnicity, and the TAPS Tool currently exists only in an English language version.

The Proposed Study: TAPS-Electronic Spanish Platform (TAPS-ESP). The current study proposes to develop a technology platform for delivering the TAPS Tool to a Spanish-speaking, health disparity population in community health centers. This Phase 1 STTR project will involve: the adaptation of the TAPS into Spanish, its development on a self-administered mobile/tablet technology platform, and an empirical study of its preliminary validity, feasibility, and acceptability in a Spanish-speaking primary care sample. The investigators refer to this novel adaptation of the TAPS Tool as the TAPS-Electronic Spanish Platform, or TAPS-ESP.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* A patient at the established clinic site
* Spanish-language dominant (with ability to read Spanish)

Exclusion Criteria:

* Unable to provide informed consent (e.g., due to acute impairment or psychosis)
* Inability to comprehend or read Spanish
* Inability to self-administer the iPad tool due to physical limitations
* Previously enrolled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Translation of the Tobacco, Alcohol, Prescription drug, and illicit Substance Use Tool (TAPS Tool) | Estimated 4 Month
  To conduct a research-driven translation and adaptation of the TAPS Tool into a Spanish-language, self-administered mobile/tablet platform (TAPS-ESP), informed by cognitive interviews with 10 Spanish-speaking primary care patients.
Preliminary Examination of the translated Tobacco, Alcohol, Prescription drug, and illicit Substance Use Tool-Electronic Spanish Platform (TAPS-ESP) | Estimated 4 Month
  To conduct a preliminary examination of the validity of the TAPS-ESP with 100 Spanish-speaking primary care patients, compared to established Spanish-language reference standard measures
Feasibility and Acceptability of the Tobacco, Alcohol, Prescription drug, and illicit Substance Use Tool-Electronic Spanish Platform (TAPS-ESP) | Estimated 4 Months
  To determine the (a) feasibility and (b) acceptability of the TAPS-ESP (including patient perspectives and preferences regarding TAPS-ESP integration with electronic health records) among Spanish-speaking adult primary care patients, using a brief survey with the 100 participants in the validation study.

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor Scott & White Research Institiute, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sanchez K, Gryczynski J, Carswell SB, Schwartz RP. Development and Feasibility of a Spanish Language Version of the Tobacco, Alcohol, Prescription Drug, and Illicit Substance Use (TAPS) Tool. J Addict Med. 2021 Jan-Feb 01;15(1):61-67. doi: 10.1097/ADM.0000000000000699. PMID 32657958